CLINICAL TRIAL: NCT00575939
Title: Assessment of the Use of a Metabolically-friendly Antiretroviral Regimen to Slow Down the Rate of Progression in Carotid Artery Intima-medial Thickness in Adults With HIV
Brief Title: Antiretrovirals and Rate of Progression in Carotid Artery Intima-medial Thickness in HIV
Status: Completed | Type: Observational
Sponsor: University Hospitals Cleveland Medical Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Grace McComsey, Professor of Pediatrics and Medicine, University Hospitals Cleveland Medical Center
Other Study IDs: AIDS 070711; BMS
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: HIV Infections; Atherosclerosis
Keywords: HIV; IMT; coronary; Treatment Naive
MeSH Terms: conditions — HIV Infections; Atherosclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stored plasma and serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HIV positive: HIV infected treatment naive with CD4 cell count of at least 400
- Healthy controls: Healthy controls

SUMMARY:
It is well known that HIV-infected subjects frequently experience hyperlipidemias, insulin resistance, and visceral adiposity, which are known to increase the risk of atherosclerosis. Several cohorts have shown an increased risk of heart disease in people with HIV. The effect of HIV treatment versus HIV itself on the incidence of heart disease is unclear. In this study the investigators will assess the effect on carotid IMT of the initiation of antiretroviral combinations that are known to have a minimal effect on lipids and insulin resistance. We will also assess the changes in several inflammation and cardiovascular markers,as well as endothelial activation markers,and how these changes relate to therapy-induced changes in immunologic, virologic and metabolic markers.

ELIGIBILITY:
Inclusion Criteria for HIV positive group:

* HIV-1 infection
* Age at least 18 years
* Naïve to antiretroviral therapy
* CD4 cell count > 400 cells/mm3

For controls: Age at least 18 years, no known HIV infection, and no known medical condition requiring chronic use of prescription medications.

Exclusion Criteria (both groups):

* Diabetes
* Pregnant or breastfeeding
* Women of child bearing age who refuse or are unable to use appropriate methods of contraception during the entire study period.
* Active infectious or inflammatory condition
* In jail or involuntarily incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 80 HIV-infected adults older than 18 years of age, ART-naïve with CD4 count of at least 400 cells/mm3
  The control group will be adults, healthy controls with no active infection or inflammatory condition, who are matched by gender and age to the HIV positive group
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2007-11; Primary Completion 2013-07 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Changes in Carotid IMT | Annualy for 4 years

SECONDARY OUTCOMES:
Increase or decrease in Inflammatory markers | Annually for 4 years
Changes in Fasting lipids | Annually for 4 years
Change in Insulin resistance by HOMA score | Annually for 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Grace A McComsey, MD, Principal Investigator — Case Western Reserve University and University Hospitals of Cleveland
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States